CLINICAL TRIAL: NCT05998200
Title: Safety of Serum Containing Alpha Hydroxy Acid (AHA) and Polyglutamate Acid Derivatives for Post-Inflammatory on Hyperpigmentation Skin
Brief Title: Safety of Serum for Post-Inflammatory on Hyperpigmentation Skin
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ungku Shahrin Medical Aesthetic Research & Innovation (USMARI) Centre (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UMRAMREC001-23
Record Dates: First submitted 2023-08-01; First posted 2023-08-18 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Healthy
Keywords: Aesthetic; Cosmetic; Post-inflammatory hyperpigmentation (PIH)
MeSH Terms: conditions — Hyperpigmentation | interventions — glycolic acid; Lactic Acid; Prostaglandins A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Serum with low concentration AHA (1% Glycolic acid and Lactic acid) and PGA (Other): This serum containing low concentration AHA (1% Glycolic acid and Lactic acid) and PGA.
  Interventions: Other: Serum with low concentration AHA (1% Glycolic acid and Lactic acid) and PGA

INTERVENTIONS:
Other: Serum with low concentration AHA (1% Glycolic acid and Lactic acid) and PGA — Participants will used the serum twice daily for 8 weeks

SUMMARY:
This study aims to investigate the safety of serum product containing low dose of alpha hydroxy acid (AHA) i.e. 1% Glycolic acid and Lactic acid and Polyglutamate acid derivatives (PGA) for post-inflammatory hyperpigmentation skin in Malaysia. The study duration is 8 weeks and the skin assessment will be carried out at baseline, week 4 and week 8.The main questions this study aims to answer are:

1. To investigate the safety of serum containing low concentration AHA (1% Glycolic acid and Lactic acid) and PGA for post-inflammatory hyperpigmentation skin among Malaysian.
2. To assess the patient satisfaction after using serum containing low concentration AHA (1% Glycolic acid and Lactic acid) and PGA among Malaysian.

ELIGIBILITY:
Inclusion Criteria:

* Malaysian from 18 to 40 years old.
* Participants with post-inflammatory hyperpigmentation (PIH).

Exclusion Criteria:

* Participant with known systemic or skin disease and any underlying medical illness
* Pregnant, breastfeeding women or planned pregnancy during the study period.
* Had reported history of dermatologic conditions (i.e. Atopic dermatitis, psoriasis) or known allergies to any ingredients that may be found in the product.
* Had any cosmetic procedures such as Botox, laser and light treatment, facial surgery, chemical peel and any procedures that may improve skin texture 1 month before the study.
* Had history of taking isotretinoin for the past 6 or 12 month and AHA (alpha hydroxyl acids) containing products or any other products for treating hyperpigmentation skin or melasma 1 month prior to study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Adverse effect after using the serum. | Week 8
  Based on adverse effect occurrence on participants that occur during study period (8 weeks)

SECONDARY OUTCOMES:
Change in skin moisture level | Baseline, Week 4 and Week 8
  Skin moisture will be measure using JANUS III skin analyzer and the changes in skin moisture from baseline and at week 4 and week 8 will be compared.
Change in skin spot level | Baseline, Week 4 and Week 8
  Skin spot will be measure using JANUS III skin analyzer and the changes in skin spot from baseline and at week 4 and week 8 will be compared.
Change in skin pores level | Baseline, Week 4 and Week 8
  Skin pores will be measure using JANUS III skin analyzer and the changes in skin pores from baseline and at week 4 and week 8 will be compared.
Change in skin tone level | Baseline, Week 4 and Week 8
  Skin tone will be measure using JANUS III skin analyzer and the changes in skin tone from baseline and at week 4 and week 8 will be compared.
Participant satisfaction after using the serum for 8 week. | Week 8
  Participation satisfaction will be evaluated using the Physician Global Assessment (PGA) survey. The subjective score of changes in skin conditions including skin wrinkles, dryness, smoothness, moisturizing and brightening effect will be graded as follows: very satisfied, satisfied, neutral, dissatisfied, very dissatisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- Ungku Shahrin Medical Aesthetic Research & Innovation (USMARI) Centre, Petaling Jaya, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No